CLINICAL TRIAL: NCT05820009
Title: Evaluation of the GORE® VIABIL® Biliary Endoprosthesis in the Treatment of Benign Biliary Strictures Secondary to Chronic Pancreatitis
Brief Title: GORE® VIABIL® Biliary Endoprosthesis in the Treatment of Benign Biliary Strictures Secondary to Chronic Pancreatitis
Acronym: VIABILITY
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The Gore VIABILITY Pivotal Study is being suspended. The suspension is not due to any safety or performance concerns. No sites have been activated and no subjects have been enrolled in the study.
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBL 22-01
Record Dates: First submitted 2023-03-16; First posted 2023-04-19 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pancreatitis, Chronic; Stricture; Bile Duct
Keywords: Benign Bile Duct Stricture
MeSH Terms: conditions — Pancreatitis, Chronic; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GORE® VIABIL® Biliary Endoprosthesis (Experimental): GORE® VIABIL® Biliary Endoprosthesis
  Interventions: Device: GORE® VIABIL® Biliary Endoprosthesis; Device: GORE® VIABIL® Short Wire Biliary Endoprosthesis

INTERVENTIONS:
Device: GORE® VIABIL® Biliary Endoprosthesis — Endoscopic treatment of benign biliary stricture secondary to Chronic Pancreatitis with the GORE® VIABIL® Biliary Endoprosthesis.
Device: GORE® VIABIL® Short Wire Biliary Endoprosthesis — Endoscopic treatment of benign biliary stricture secondary to Chronic Pancreatitis with GORE® VIABIL® Short Wire Biliary Endoprosthesis

SUMMARY:
This study will evaluate the safety and effectiveness of the GORE® VIABIL® Biliary Endoprosthesis in the treatment of benign biliary strictures secondary to Chronic Pancreatitis (CP).

DETAILED DESCRIPTION:
A maximum of 15 clinical investigative sites across the U.S. will participate in this study. One hundred and thirty-three subjects are intended to be implanted with the GORE® VIABIL® Biliary Endoprosthesis in this study. Subjects will be evaluated at the time of device placement and will have follow-up visits at 1 week and 1, 3, 6, and 9 months during indwell; subjects will have the device removed at 10-12 months and have post removal follow-up visits at 1 week and 1, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria

1. A diagnosis of chronic pancreatitis
2. Indication for ERCP with FCSEMS placement determined by one or more of the following:

   1. Presence of a Bismuth type I BBS confirmed by imaging (e.g., cholangiography, Computed Tomography [CT], Magnetic Resonance Cholangiopancreatography [MRCP], etc.) collected ≤ 60 days prior to the index procedure and an elevation of serum alkaline phosphatase (>2 times the upper limit of institutional reference range)
   2. Presence of a symptomatic (e.g., jaundice, cholangitis, and/or choledocholithiasis) Bismuth type I BBS confirmed by imaging (e.g., cholangiography, CT, MRCP, etc.) collected ≤ 60 days prior to the index procedure with an elevation of serum alkaline phosphatase (>2 times the upper limit of institutional reference range)
   3. A planned exchange of multiple side-by-side plastic stents (whose combined diameters are ≤ 20 Fr) that were previously placed for management of a Bismuth type I BBS secondary to chronic pancreatitis
3. Underlying stricture malignancy has been reasonably excluded (e.g., by any of the following techniques - biopsy, Endoscopic Ultrasound [EUS], Computed Tomography [CT], or Magnetic Resonance Imaging [MRI] with or without Magnetic Resonance Cholangiopancreatography [MRCP]) ≤ 60 days prior to index procedure
4. ≥ 18 years old at the time of informed consent signature
5. Male, infertile female, or woman of childbearing potential with a negative beta Human Chorionic Gonadotropin (hCG) pregnancy test within 7 days of the index procedure
6. Able and willing to provide written informed consent (or has a Legally Authorized Representative) to participate in the study prior to any study procedures
7. Willing and able to comply with the study procedures and follow-up requirements

Exclusion Criteria

1. Concurrent participation in another interventional study that involves an investigational product being introduced to the body
2. A contraindication for endoscopic techniques
3. Life expectancy < 2 years
4. A history of malignant biliary or malignant pancreatic disease
5. Prior or existing biliary self-expanding metal stent (SEMS)
6. Prior or planned exchange of multiple side-by-side plastic stents whose combined diameters are greater than 20 Fr
7. Development of obstructive biliary symptoms associated with a present attack of acute pancreatitis
8. Any biliary stricture etiology other than chronic pancreatitis
9. Other therapeutic endoscopic procedures performed during the index or removal procedure that are not associated with bile duct stricture secondary to Chronic Pancreatitis including but not limited to planned Fine Needle Aspiration (FNA) or Fine Needle Biopsy (FNB) of the pancreas
10. Concomitant Bismuth type II-IV stricture
11. Inability for the guidewire to traverse the papillae and the stricture (e.g., as a result of surgically altered anatomy)
12. Inability to pass the endoscope to the papillae without the need for mechanical dilation
13. Known bile duct fistula or leak
14. Biliary stricture length > 100 mm (10 cm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Safe stent removal as reported by serious adverse event reporting | At removal (10-12 months)
  Ability to remove the Study Device endoscopically without stent removal-related serious adverse events (SAEs) as assessed from the time of Study Device removal to one month (30 days) post-Study Device removal.

SECONDARY OUTCOMES:
Placement success as determined by imaging | Day 0
  Ability to deploy the Study Device in a satisfactory position across the biliary stricture.
Stent functionality as determined by adverse event reporting | During indwell up to 12 months
  Defined as freedom from Study Device-related reintervention during intended indwell
Migration as determined by imaging | During indwell up to 12 months
  Defined as movement of the Study Device such that the Study Device is no longer in a satisfactory position across the biliary stricture during intended indwell.
Removal success as determined by imaging | At removal (10-12 months)
  Defined as either ability to remove the Study Device endoscopically at scheduled Study Device removal without stent removal-related SAEs or spontaneous Study Device passage without the need for immediate re-stenting
Stricture resolution at stent removal as determined by imaging | At removal (10-12 months)
  Defined as freedom from recurrent stent placement at the end of indwell
Stricture recurrence as determined by adverse event reporting | From removal up to 24 months
  Defined as any biliary stricture-related re-intervention from the removal procedure through 2 years post-Study Device removal.
Device- or procedure-related SAEs as determined by serious adverse event reporting | Day 0-13 months (including through 30 days post-removal)
  Defined as Study Device- or procedure-related SAEs that occur during placement, indwell, or removal (including through 30 days post-removal).
Liver Function as determined by alkaline phosphatase, alanine aminotransferase, and aspartate aminotransferase levels | Baseline, indwell follow-up visits (up to 12 months), at removal (10-12 months), and post-removal follow up visits (up to 24 months)
  Including alkaline phosphatase (ALP, U/L), alanine aminotransferase (ALT, U/L), aspartate aminotransferase (AST, U/L) levels
Liver Function as determined by direct bilirubin, and total bilirubin | Baseline, indwell follow-up visits (up to 12 months), at removal (10-12 months), and post-removal follow up visits (up to 24 months)
  Including direct bilirubin (mg/dL), and total bilirubin (mg/dL) levels

CONTACTS AND LOCATIONS:
Overall Officials: Todd Baron, MD, Principal Investigator — University of North Carolina Medical Center; Shayan Irani, MD, Principal Investigator — Virginia Mason Medical Center
Locations (2):
- United States (2):
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No